CLINICAL TRIAL: NCT00000418
Title: Psychosocial Intervention for Acute Low Back Pain (ALBP)
Brief Title: Psychosocial Treatment for Acute Low Back Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P60 AR20582 Substudy EEHSR4; P60AR020582 (NIH); NIAMS-025
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2013-06-06 (Estimated); Status verified 1999-06

CONDITIONS: Acute Low Back Pain
Keywords: OA; Patient education; Acute low back pain (ALBP); Social support systems
MeSH Terms: interventions — Psychosocial Intervention

INTERVENTIONS:
Procedure: Psychosocial intervention

SUMMARY:
Acute low back pain (severe pain that comes on suddenly and lasts a relatively short time) is very common in the United States, and accounts for substantial illness, functional limitations, pain, and health care costs. This study looks at whether a program designed to improve self-efficacy (a person's belief in his or her ability to reach a goal, such as managing one's own disease) and social support improves the health status of people with acute low back pain.

DETAILED DESCRIPTION:
Acute low back pain (ALBP) is very prevalent in the United States, accounting for substantial morbidity, functional limitations, pain, and health care costs. Psychosocial interventions that target improved symptom control and patient functioning have the potential to improve the outcomes of patients with ALBP. This study evaluates a psychosocial intervention designed to enhance self-efficacy and social support for patients with ALBP.

In this randomized, controlled trial, we will randomize eligible patients with ALBP to receive the intervention or usual care. The intervention program consists of: (1) patient education regarding ALBP; (2) explanations and rationales, in layperson's terms, of diagnostic and treatment options for ALBP; (3) discussions regarding the management of negative affect (i.e., depression, anger, fear, hostility, anxiety); (4) methods to involve social support systems; and (5) strategies to involve the primary care physician to reinforce patients' behaviors and progress. We will follow patients for 12 months and assess outcomes at 3 and 12 months.

Primary outcomes are health-related quality of life (i.e., functional status, role function, back pain symptoms) and patient satisfaction with care. Secondary outcomes include health care use, direct health care costs, self-efficacy, and social support. We will also estimate the cost-effectiveness of the intervention.

We will conduct this investigation among socioeconomically vulnerable patients with ALBP, a group that shoulders a disproportionate burden of disability and morbidity from musculoskeletal conditions and comorbid medical conditions.

ELIGIBILITY:
Inclusion Criteria:

* Acute low back pain

Exclusion Criteria:

* Chronic back pain (including surgery)
* Disability claim for back pain
* Nursing home resident
* Severe impairment in hearing, vision, or speech
* Unable to speak English
* Severe comorbidity
* Unable to contact by phone
* Excluded by primary care physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211
Dates: Start 1977-09; Study Completion 2001-03

CONTACTS AND LOCATIONS:
Overall Officials: Morris Weinberger, Ph.D., Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States

REFERENCES:
- [Background] Damush TM, Weinberger M, Clark DO, Tierney WM, Rao JK, Perkins SM, Verel K. Acute low back pain self-management intervention for urban primary care patients: rationale, design, and predictors of participation. Arthritis Rheum. 2002 Aug;47(4):372-9. doi: 10.1002/art.10382. PMID 12209482
- [Background] Damush TM, Weinberger M, Perkins SM, Rao JK, Tierney WM, Qi R, Clark DO. Randomized trial of a self-management program for primary care patients with acute low back pain: short-term effects. Arthritis Rheum. 2003 Apr 15;49(2):179-86. doi: 10.1002/art.10995. PMID 12687508
- [Background] Damush, Weinberger, Perkins, Rao, Tierney, Qi, & Clark. The cost-effectiveness of a self-management program for primary care patients with acute low back pain. 2002. In preparation.
- [Background] Damush TM, Weinberger M, Tierney WM, Rao JK, Clark DO, & Perkins SM. A randomized trial of a self-management program for primary care patients with acute low back pain: 12-month outcomes. Poster presented at the annual meeting of the American College of Rheumatology, San Francisco, CA. Arthritis & Rheumatism. 2001;44:S206.
- [Background] Damush TM, Weinberger M, Tierney WM, Rao JK, Clark DO, & Perkins SM. A randomized trial of a self-management program for primary care patients with acute low back pain: 4-month outcomes. Poster presented at the annual meeting of the American College of Rheumatology, Philadelphia, PA. Arthritis & Rheumatism. 2000;43:S9.
- [Background] Damush TM, Weinberger M, Tierney WM, Rao J, Clark DO, Adams K, Perkins S, & Emsley C. A comparison between older and younger adults with acute low back pain on functional status and self-management. Poster presented at the annual meeting of the Gerontological Society of America, San Francisco, CA. The Gerontologist. 1999;39:S571.
- [Background] Damush TM, Weinberger M, Perkins SM, Rao JK, Tierney WM, Qi R, Clark DO. The long-term effects of a self-management program for inner-city primary care patients with acute low back pain. Arch Intern Med. 2003 Nov 24;163(21):2632-8. doi: 10.1001/archinte.163.21.2632. PMID 14638564
- [Derived] Gameza VA, Bell Lybecker M, Wara P. Laparoscopic Keyhole Versus Sugarbaker Repair in Parastomal Hernia: A Long-Term Case-Controlled Prospective Study of Consecutive Patients. J Laparoendosc Adv Surg Tech A. 2020 Jul;30(7):783-789. doi: 10.1089/lap.2020.0074. Epub 2020 Mar 27. PMID 32216697